CLINICAL TRIAL: NCT00541073
Title: Phase 2 Pharmacological Study of Pemetrexed Administered With Cisplatin and a Vitamin Supplement in Patients With Nonresectable Pleural Mesothelioma
Brief Title: Pemetrexed, Cisplatin, and Vitamin B12 in Treating Patients With Mesothelioma of the Chest That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000564058; COL-ALIMESO; INCA-RECF0441; COL-2006-04
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2009-07

CONDITIONS: Malignant Mesothelioma
Keywords: advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Vitamin B 12; Cisplatin; Pemetrexed; Gene Expression Profiling

INTERVENTIONS:
Dietary Supplement: vitamin B12
Drug: cisplatin
Drug: pemetrexed disodium
Genetic: gene expression analysis
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving pemetrexed together with cisplatin and vitamin B12 may kill more tumor cells.

PURPOSE: This phase II clinical trial is studying how well giving pemetrexed together with cisplatin and vitamin B12 works in treating patients with mesothelioma of the chest that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Define an individually adapted (by dosage) protocol of pemetrexed disodium, cisplatin, and vitamin B12 in patients with unresectable pleural mesothelioma.

Secondary

* Determine the relationship between pharmacokinetic and pharmacodynamic parameters (hematologic and nonhematologic).
* Analyze the inter-individual pharmacokinetic variations and the influence of the covariables on the pharmacokinetics of pemetrexed disodium.
* Analyze the impact of pharmacogenetic (MTHFR, TS, GSTpi, ERCC1, XPD) variations on the toxicity of pemetrexed disodium.
* Validate a strategy of adapting dosage.

OUTLINE: This is a multicenter study.

Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 2 hours on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive vitamin B12 intramuscularly on day -7 and then every 9 weeks until chemotherapy is completed.

Blood samples are collected during the first and third courses of chemotherapy. Samples are analyzed by pharmacogenetic (MTHFR, TS, GSTpi, ERCC1, xPD), pharmacokinetic, and other pharmacological methods.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed pleural mesothelioma

  * Unresectable disease

Exclusion criteria:

* Clinically detected pleural effusion or ascites that cannot be controlled by drainage or other procedures

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-2
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine clearance > 45 mL/min
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Transaminases ≤ 3 times ULN (5 times ULN if liver metastases)
* Not pregnant or nursing
* Fertile patients of must use effective contraception during and for 6 months after completion of study treatment

Exclusion criteria:

* Hypersensitivity to pemetrexed disodium or any of its excipients
* Peripheral neuropathy ≥ grade 2
* Impossible to receive study therapy due to geographical, social, familial, or psychological reasons

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* At least 28 days since prior radiotherapy (21 days for injected radiotherapy)

Exclusion criteria:

* Prior chemotherapy
* Prior yellow fever vaccine
* Inability to discontinue aspirin (> 1.3 g/day) or NSAIDs for 2 days prior to, during, and 2 days after day 1 of each course of study therapy
* Concurrent participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Individual dosage-adapted protocol

SECONDARY OUTCOMES:
Relationship between pharmacokinetic and pharmacodynamic parameters
Pharmacokinetics
Pharmacogenetic variations (MTHFR, TS, GSTpi, ERCC1, XPD)

CONTACTS AND LOCATIONS:
Overall Officials: Amelie Lansiaux, MD, PhD — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France